CLINICAL TRIAL: NCT03452332
Title: Phase I Multi-Center Study of Hypofractionated Radiotherapy in Combination With Durvalumab and Tremelimumab in Patients With Recurrent/Metastatic Advanced Cervical, Vaginal, or Vulvar Cancer
Brief Title: Stereotactic Body Radiation Therapy, Tremelimumab and Durvalumab in Treating Participants With Recurrent or Metastatic Cervical, Vaginal, or Vulvar Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0548; NCI-2018-00627 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0548 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Advanced Cervical Adenocarcinoma; Advanced Vaginal Carcinoma; Advanced Vulvar Carcinoma; Human Papillomavirus-Related Cervical Squamous Cell Carcinoma; Human Papillomavirus-Related Vulvar Squamous Cell Carcinoma; Metastatic Cervical Adenocarcinoma; Metastatic Cervical Carcinoma; Metastatic Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Metastatic Vaginal Adenocarcinoma; Metastatic Vaginal Carcinoma; Metastatic Vulvar Carcinoma; Recurrent Cervical Adenocarcinoma; Recurrent Cervical Carcinoma; Recurrent Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Recurrent Vaginal Carcinoma; Recurrent Vulvar Carcinoma; Stage III Cervical Cancer AJCC v8; Stage III Vaginal Cancer AJCC v8; Stage III Vulvar Cancer AJCC v8; Stage IIIA Cervical Cancer AJCC v8; Stage IIIA Vulvar Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IIIB Vulvar Cancer AJCC v8; Stage IIIC Vulvar Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Vaginal Cancer AJCC v8; Stage IV Vulvar Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Vaginal Cancer AJCC v8; Stage IVA Vulvar Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8; Stage IVB Vaginal Cancer AJCC v8; Stage IVB Vulvar Cancer AJCC v8; Vaginal Squamous Cell Carcinoma, Not Otherwise Specified; Vulvar Adenocarcinoma; Vulvar Squamous Cell Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; Radiosurgery; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tremelimumab, durvalumab, SABR) (Experimental): Participants receive tremelimumab IV over 1 hour followed by durvalumab IV over 1 hour on day 1 of each cycle. Participants also undergo SABR over 30-45 minutes on days 8, 10, and 12 of cycle 1. Treatment with tremelimumab repeats every 4 weeks for up to 4 cycles, and treatment with durvalumab repeats every 4 weeks for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Radiation: Stereotactic Radiosurgery; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Stereotactic Radiosurgery — Undergo SABR
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
This phase I trial studies how well stereotactic body radiation therapy works in combination with tremelimumab and durvalumab in treating participants with cervical, vaginal, or vulvar cancers that have come back (recurrent) or spread to other areas of the body (metastatic). Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue. Immunotherapy with monoclonal antibodies, such as tremelimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Durvalumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Giving stereotactic body radiation therapy, tremelimumab, and durvalumab may work better in treating participants with cervical, vaginal, or vulvar cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, and tolerability of combined immune checkpoint blockade with 3 fractions of stereotactic body radiation therapy (stereotactic ablative radiotherapy [SABR]) of up to two metastatic lesions in patients with recurrent and or metastatic cervical, vaginal, or vulvar cancer.

SECONDARY OBJECTIVES:

I. To evaluate clinical response rates and assess toxicities of treatment to durvalumab combined with tremelimumab with 3 fractions of SABR of at least one and up to two metastatic lesions in patients with recurrent/metastatic cervical, vaginal, or vulvar cancer.

II. To estimate progression-free survival, overall survival, and time to next treatment.

EXPLORATORY OBJECTIVES:

I. To evaluate potential biomarkers of immune response to combined immune-checkpoint inhibition with SABR and correlate this with clinical response to treatment.

II. To evaluate potential biomarkers of immune response including cervical and rectal microbial diversity, cervical immune cell infiltration and peripheral immune cell activation as correlates of clinical response to treatment.

OUTLINE:

Participants receive tremelimumab intravenously (IV) over 1 hour followed by durvalumab IV over 1 hour on day 1 of each cycle. Participants also undergo SABR over 30-45 minutes on days 8, 10, and 12 of cycle 1. Treatment with tremelimumab repeats every 4 weeks for up to 4 cycles, and treatment with durvalumab repeats every 4 weeks for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days, at 2, 3, 4, 6, 8, 10, and 12 months, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from subject prior to any protocol related procedures
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2.
* Body weight > 30 kg
* Must have an average life expectancy of 6 months
* Patient is able and willing to comply with protocol and study procedures for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up visits
* Histological diagnosis of recurrent or metastatic cervical, vaginal, or vulvar cancer or an unknown pelvic malignancy most likely to have arisen from these sites as determined clinically by the treating physicians (i.e. squamous cell carcinoma or adenocarcinoma that is high risk [HR] human papillomavirus positive [HPV]+, but not limited to this example)
* Metastatic disease in at least two distinct lesions (including the index lesion to be treated) with at least one site outside of the radiation field and evaluable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria for evaluation of response
* At least one index lesion to be treated measuring 1 cm amenable to hypofractionated radiation therapy
* Staging computed tomography (CT) scans done prior to enrollment
* Have had at least one line of prior platinum-based systemic chemotherapy once diagnosed with recurrence or metastatic disease if primary cervical cancer. If a patient has primary vulvar or vaginal cancer, there is not a requirement.
* May have received 1 prior biologic regimen (i.e. avastin) but not within 4 weeks of enrollment
* Full recovery from the acute effects of prior treatments, defined as effects having resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03 grade 0 or 1 with the exception of alopecia and certain laboratory values as outlined below; subjects with irreversible toxicity that is not reasonably expected to be exacerbated by durvalumab and tremelimumab may be included (e.g., hearing loss, neuropathy) upon approval of the principal investigator (PI)
* In patients with central nervous system (CNS) metastases, metastases must be asymptomatic at the time of day 1 of the study and meet the following criteria:

  * Brain metastases should have been treated with either whole brain radiation therapy (WBRT), stereotactic radiosurgery (SRS)/gamma-knife, or surgical resection;
  * At least 28 days without progression of CNS metastases as evidenced by magnetic resonance imaging (MRI) or CT from last day of treatment with radiation to the CNS metastases;
  * At least 3 months from surgical resection (if had surgery) with stability on MRI brain at enrollment;
  * At least 14 days since last dose of corticosteroids;
  * Must not have leptomeningeal disease or cord compression
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN); for subjects with liver metastasis, ALT and AST =< 5 x ULN within 3 weeks prior to initial treatment
* Total bilirubin =< 1.5 x ULN except in patients with documented Gilbert's syndrome or liver metastasis, who must have a baseline total bilirubin =< 3.0 mg/dl within 3 weeks prior to initial treatment
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance within 3 weeks prior to initial treatment
* Negative screening test results for hepatitis B, hepatitis C, and human immunodeficiency virus
* Absolute neutrophil count (ANC) >= 1,500 cells/ul without growth factor support prior to initial treatment
* Hemoglobin >= 9 g/dL prior to initial treatment
* Platelet count >= 100,000 platelets/ul prior to initial treatment
* Subjects must either be of non-reproductive potential (ie, post-menopausal by history; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum or urine pregnancy test upon study entry; women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause; the following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy); they would also be considered had radiation-induced or chemotherapy-induced menopause with last menses > 1 year ago
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
  * Women of any age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced or chemotherapy-induced menopause
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use highly effective method of contraception from the time of screening, and must agree to continue using such precautions for 180 days after the final dose of durvalumab and tremelimumab; cessation of contraception after this point should be discussed with a responsible physician; they must also refrain from egg cell donation for 180 days after the final dose of durvalumab and tremelimumab

  * Note: A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly; the acceptable methods of contraception include barrier methods (male condom plus spermicide, copper T intrauterine device, levonorgesterel-releasing intrauterine system) or hormonal methods (implants, hormone shot or injection, combined pill, minipill, patch)

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Previous enrollment in the present study
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy
* Prior treatment with an anti-CTLA-4, including tremelimumab PD-1 or PD-L1 inhibitor, including durvalumab
* Prior oncology vaccine therapy
* Prior radiation treatment to the index lesion to be treated
* Prior radiation which overlaps and precludes hypofractionated treatment to the index lesion
* Treatment with other investigational agent within 4 weeks to the first dose of tremelimumab or durvalumab
* Concomitant therapy with any of the following: interleukin-2 (IL-2), interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; all such therapies must have been discontinued > 4 weeks
* Any unresolved toxicity (CTCAE grade < 2) from previous anti-cancer therapy; (subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
* Any prior grade >= 3 immune-related adverse event (imAE) while receiving any previous immunotherapy agent, or any unresolved imAE > grade 1
* Treatment with a vascular endothelial growth factor (VEGF) inhibitor within the last 6 weeks
* Major surgical procedure (as defined by the treating physician) within 28 days prior to the first dose of durvalumab and tremelimumab or still recovering from prior surgery
* Active cardiac disease defined as unstable angina, uncontrolled hypertension, myocardial infarction in the last six months (unless successfully treated with coronary artery bypass grafting [CABG] or percutaneous transluminal coronary angioplasty [PTCA]), uncontrolled arrhythmia, or symptomatic congestive heart failure; > 3 heart-related hospitalizations in the past year
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from 3 electrocardiogram (ECGs) using Fridericia's correction from triplicate ECGs in those patients who have an initial abnormal EKG on screening
* Severe chronic obstructive pulmonary disease (COPD) requiring > 3 hospitalizations in the past year
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]); the following are exceptions to this criterion:

  * Patients with vitiligo or alopecia;
  * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement;
  * Any chronic skin condition that does not require systemic therapy;
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician;
  * Patients with celiac disease controlled by diet alone
* Active or prior documented interstitial lung disease
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab and tremelimumab with the exceptions of intranasal and inhaled corticosteroids, systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent, or steroids used transiently to control contrast agent allergies for radiographic studies
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or tremelimumab or any CTLA4, PD1, or PDL-1 inhibitor
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies); patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible; patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* History of prior bowel fistula, ulcerations, or perforations
* Evidence of progressive or symptomatic central nervous system (CNS) metastases or leptomeningeal disease
* Uncontrolled inter-current illness, including, but not limited to, ongoing or active infection requiring systemic treatment, current or history of prior radiation induced pneumonitis, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement or compromise the ability of the subject to give written informed consent
* Other active invasive malignancy; history of non-invasive malignancies such as ductal carcinoma in situ of the breast, non-melanomatous carcinoma of the skin, is allowed, as is history of other invasive malignancy that is in remission for >= 5 years after treatment with curative intent
* Any medical, psychological, or social condition that, in the opinion of the treating physician would interfere with evaluation of the investigational product or interpretation of subject safety or study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03 | Up to 3 months after last dose of durvalumab
  Will be assessed based on dose limiting toxicities (DLTs) and based on adverse events (AEs) throughout the entire treatment period. In the overall assessment of adverse events, AEs will be tabulated by body system, type and grade, overall and by disease cohort. The number and percentage of patients experiencing at least one grade 3 or higher AE will also be reported.

SECONDARY OUTCOMES:
Response to treatment by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and immune-related response criteria | Up to 1 year
  This will be measured in both treated and untreated lesions with computed tomography (CT) imaging or other appropriate imaging modalities. Immune-related response is reported as number and percent of patients with two-sided 80% confidence intervals (CI). Because each patient will have multiple lesions, a generalized linear mixed model will be used, if possible, to calculate overall response, as well as response by index or non-index lesion. The depth and duration of response will be depicted using waterfall and swimmer plots.
Progression-Free Survival | From the start of therapy up to first documented disease progression or death from any cause, assessed up to 1 year
  To summarize progression free survival we will use Kaplan Meier analysis, reporting the median with confidence interval.
Overall Survival | From start of therapy to death from any cause, assessed up to 1 year
  To summarize overall survival we will use Kaplan Meier analysis, reporting the median with confidence interval.
Time to next treatment (TTNT) | From the end of immune-checkpoint inhibition treatment to institution of next therapy, assessed up to 1 year
  To summarize time to next treatment we will use Kaplan Meier analysis, reporting the median with confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Lilie L Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org